CLINICAL TRIAL: NCT05527353
Title: Human Anti-MülleRian Hormone for Diagnosis of PCOS Study
Brief Title: AMH for the Identification of PCOM in PCOS Diagnosis
Acronym: HARMONIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oulu University Hospital (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 49/2019
Record Dates: First submitted 2022-08-05; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; PCOS; anti-müllerian hormone; AMH; antral follicle count; polycystic ovarian morphology
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with PCOS: Women born in Northern Finland during 1985-1987 fulfilling ≥2 Rotterdam criteria.
- Controls: Women born in Northern Finland during 1985-1987 who are PCOM negative with no other diagnostic features of PCOS according to the Rotterdam criteria.

SUMMARY:
The purpose of this study is to validate the anti-müllerian hormone (AMH) cut-off established and validated in the APHRODITE study, for the determination of PCOM as part of the diagnosis of PCOS, using the Elecsys AMH Plus immunoassay.

DETAILED DESCRIPTION:
The study participants will be women born July 1985-Dec 1987 in Northern Finland; the study partially links to the Northern Finland Birth Cohort 1986. Female subjects included in this cohort will be invited to participate in the study with the aim to enroll up to 1800 subjects. Each enrolled subject will have one study visit, where the clinical data required for assessing their PCOS status will be recorded, including a gynecological examination by transvaginal ultrasound to determine polycystic ovarian morphology (PCOM) status (antral follicle count and ovarian volume). Study subjects will also have blood drawn for serum collection, where hormonal parameters relevant for PCOS will be measured. The collected serum will also be used to measure the AMH levels using the Roche Elecsys AMH test.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Born July 1985-Dec 1987 in Northern Finland
* Signed informed consent regarding ROCHE collaboration

Exclusion Criteria:

* Unwilling to undergo gynecological examination including transvaginal ultrasound (TVUS)
* Unwilling to have blood drawn
* Pregnancy

Ages: 32 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Subjects born in Northern Finland in July 1985- December 1987 who were assigned female at birth and currently register as females.
Study Population: As the study is population-based, all non-pregnant women born in Northern Finland between July 1985-December 1987 will be invited to participate in the study. Most women will be white with a small minority (estimated below 3%) of indigenous Sámi people.
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The validation of the performance of the AMH cut-off, established in the APHRODITE study, to diagnose PCOM in the context of PCOS diagnosis. | Baseline
  The performance (sensitivity and specificity) of the AMH cut-off will be calculated by comparing the AMH values to the PCOM status of the subjects based on the TVUS findings (AFC & Ovarian volume).

SECONDARY OUTCOMES:
Prevalence of PCOS in general population | Baseline
  PCOS is diagnosed based on the Rotterdam Criteria with the presence of at least two of the following symptoms: 1. Polycystic ovarian morphology by trans-vaginal ultrasound (>=20 follicles in either ovary or ovarian volume >= 10 mL), 2. Hyperandrogenism, either clinical or biochemical (testosterone/free androgen index) and 3. oligo-amenorrhea (< 8 menstruations/year).

CONTACTS AND LOCATIONS:
Overall Officials: Terhi T Piltonen, Professor, Principal Investigator — Oulu University Hospital, University of Oulu
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited into the Arctic Biobank as part of the Northern Finland Birth Cohort 1986 data.
Time Frame: Data is available on request 10 years from study completion
Access Criteria: Data available according to policies of the NFBC.
URL: https://www.oulu.fi/en/university/faculties-and-units/faculty-medicine/northern-finland-birth-cohorts-and-arctic-biobank/nfbc-aineistopyynto

REFERENCES:
- [Derived] Piltonen TT, Kinnunen J, Komsi E, Kangasniemi MH, Luiro K, Rajecki M, Jokelainen J, Kiviniemi E, Allegranza D, Hund M, Olziersky AM, Logan CA, Buck K, Savukoski SM, Arffman RK. Prospective validation of anti-Mullerian hormone cutoff to determine polycystic ovarian morphology: HARMONIA study. Fertil Steril. 2025 Sep;124(3):543-552. doi: 10.1016/j.fertnstert.2025.05.147. Epub 2025 May 19. PMID 40398715
- [Derived] Piltonen TT, Allegranza D, Hund M, Buck K, Sillman J, Arffman RK. Validation of an Anti-Mullerian Hormone Cutoff for Polycystic Ovarian Morphology in the Diagnosis of Polycystic Ovary Syndrome in the HARMONIA Study: Protocol for a Prospective, Noninterventional Study. JMIR Res Protoc. 2024 Feb 6;13:e48854. doi: 10.2196/48854. PMID 38319689